CLINICAL TRIAL: NCT01310374
Title: Humoral and Cellular Immune Response Study of Influenza Vaccine
Brief Title: Immune Response Study of Influenza Vaccine
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Wu Jiang, Centers for Disease Control and Prevention, China, Centers for Disease Control and Prevention, China
Other Study IDs: BJCDCWJ201101
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Influenza Vaccine Allergy; Cell Mediated Reaction
Keywords: influenza vaccine; immune response; dynamic changes
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
An observational clinical study will be performed in subjects aged 12-60 years old to describe the dynamic changes of humoral immune/cellular immunity after vaccination of influenza vaccine, and to discuss the role of different antibodies against influenza virus infection, and to look for possible factors related to side effects with the vaccine.

DETAILED DESCRIPTION:
A randomized clinical trial will be conducted to describe immune response of seasonal influenza virus vaccine in a single center in China. 200 subjects aged 18-60 years will be enrolled under the premise of informed consent and receive one dose of vaccine. All vaccinations will be done by specific study personnel, who do not take part in the assessment of safety or immunogenicity. Adverse events will be recorded after vaccination and blood samples were collected at 0,7,14,28 days for antibody detection and split vaccine neutralizing antibody detection, determination of cellular immune function in the same time.

The clinical program approved by the ethics committee will be performed by the researchers independently. Inspectors designated by the sponsor will take meticulous on-site audits to ensure the safety specifications during the whole process of research.

ELIGIBILITY:
Inclusion Criteria:

* aged 12-60 years old
* male or non-pregnant female
* volunteers
* clinically healthy as determined by: medical history inquiring and physical examination
* provide written informed consents before joining the trial

Exclusion Criteria:

* infected with Influenza A virus subtype H1N1(2009),
* vaccinated with seasonal influenza vaccine,
* allergic to any ingredient of vaccine,
* autoimmune disease or immunodeficiency,
* active malignancy,
* bleeding disorder,
* seizure disorder,
* Guillain-Barre Syndrome,
* treatment with cytotoxic or immunosuppressive drugs within the past 6 months,
* receipt of blood products within the past 3 months,
* administration of any other investigational research agents or live attenuated vaccine within 30 days,
* administration of subunit or inactivated vaccines within 14 days,
* axillary temperature over 37.0℃ at the time of vaccination.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the dynamic changes of humoral immune/cellular immunity after vaccination of influenza vaccine | one year

CONTACTS AND LOCATIONS:
Overall Officials: jiang wu, Bachelor, Principal Investigator — Beijing Centers for Disease Control and Prevention